CLINICAL TRIAL: NCT05375409
Title: Cognitive Compensation Mechanism in the Postoperative Delirium
Brief Title: Evidence for Cognitive Compensation Mechanism in the Postoperative Delirium: a Prospective Multi-modal Neuroimaging Cohort Study in Patients With Frontal Glioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Guobin Zhang
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Delirium
Keywords: postoperative delirium; multi-model imaging
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Postoperative Delirium (+)
- Postoperative Delirium (-)
- Healthy Control

SUMMARY:
In this study, patients with frontal glioma will be selected for preoperative neurocognitive assessment, APOE genotype detection, 3D structural imaging, cortical blood oxygen level dependent imaging (resting state + task state), and subcortical diffusion tensor multimodal MRI to explore preoperative brain structures and brain networks, and postoperative delirium will be assessed 1-3 days after surgery. The aim was to investigate the preoperative neuroanatomical basis of postoperative delirium in this population at the level of brain structure and network connectivity, and to predict the risk of patients by integrating cognitive indicators and neuroimaging markers in an event probability model to construct an optimal sequence of abnormalities in a series of markers, and then to establish a more population-specific subgroup prediction based on different APOE genotypes and the establishment of neurological compensation. The final clinical validation was performed on a small sample to provide a basis for the prevention of postoperative delirium in frontal glioma patients.

DETAILED DESCRIPTION:
Delirium is an acute, reversible, widespread alteration of cognitive function characterized by fluctuating cognitive dysfunction, decreased level of consciousness, inattention, disorganized thinking, or disturbed sleep-wake cycles. Postoperative delirium is a common postoperative complication in surgical patients, occurring 1-3 days after surgery and fluctuating between 11-51% depending on the patient's age, type of surgery, and preoperative underlying disease. Postoperative delirium significantly increases perioperative complications and mortality and may leave severe long-term cognitive impairment. However, there is a relative lack of studies addressing delirium after neurosurgical craniotomy. This population may be at high risk for postoperative delirium given the direct impact of intracranial primary lesions on brain structure and function. Our team has completed a prospective cohort study (registry number: NCT03087838) enrolling 800 post-neurosurgical craniotomy patients and found for the first time that patients with gliomas had the highest incidence of postoperative delirium relative to other intracranial occupying lesions at 37.7%, especially frontal gliomas at 53.3%, and that the incidence of delirium was much higher in patients with high-grade gliomas than in patients with low The incidence of delirium was much higher in patients with high-grade gliomas than in patients with low-grade gliomas (50% vs. 16.7%) (the results of the study have not yet been published). Why is the incidence of postoperative delirium higher in patients with gliomas, especially frontal gliomas, than in other lesions, given that they are intracranial occurrences? This question caused us to think about it.

Glioma is the most common intracranial malignancy, accounting for approximately 80% of malignant brain tumors. Recent studies have found that neurocognitive dysfunction is a more common phenomenon in glioma patients and is closely associated with a decrease in health-related quality of life (HRQOL) in patients. Therefore, as the level of glioma treatment improves, patient survival is prolonged, and quality of life is increasingly emphasized, neurocognitive dysfunction has become a hot issue in the field of glioma. Postoperative delirium, as a clear and important "catalyst" for postoperative cognitive dysfunction, deserves more attention.

Given that the treatment of delirium is uncertain and that 30-40% of postoperative delirium is preventable, it is important to screen for high-risk groups. This project will explore the neuroanatomical basis of postoperative delirium in frontal glioma patients using multimodal magnetic resonance technology preoperatively, and integrate neuroimaging features and cognitive events with multidimensional clinical neurocognitive assessment to construct and validate a risk assessment model to predict postoperative delirium in this population. The significance of this study is: (1) to investigate the pathogenesis of postoperative delirium in frontal glioma patients, to explore the objective neuroimaging features with high specificity and sensitivity in vivo, and to provide new ideas and methods for the pathophysiological mechanisms of postoperative delirium; (2) the construction of the prediction model may help to provide early warning of postoperative delirium in glioma patients, which is of great clinical significance for perioperative management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with frontal glioma as revealed by head MRI, aged 18-60 years, with no history of serious disease, and who signed an informed consent form were included in the study. Controls were healthy volunteers of the same age group used for functional MRI resting state data control.

Exclusion Criteria:

* (1) patients who cannot cooperate with preoperative neurocognitive assessment and preoperative functional MRI; (2) patients with psychiatric disorders; (3) patients with a history of hydrocephalus, cerebral infarction, or cerebral hemorrhage; (4) patients with epilepsy and a history of antiepileptic drugs; (5) patients who have taken sedative or analgesic drugs within 24 hours of study entry; (6) patients with drug and alcohol abuse; (7) patients with perinatal and lactating conditions; (8) patients with recurrent intracranial tumors; (9) patients with multiple intracranial tumors; (10) patients who have undergone surgery for radiation or chemotherapy; (11) patients with multiple intracranial tumors. (6) patients with drug and alcohol abuse; (7) perinatal and lactating patients; (8) patients with recurrent intracranial tumors; (9) patients with multiple intracranial tumors; (10) patients who have undergone surgery with radiotherapy or chemotherapy; (10) patients with claustrophobia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with frontal glioma on MRI of the head, age 18-60 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
occurrance of postoperative delirium | 1-3day after surgery
  POD(+) POD(-)
preoperative cognitive examination | before sugery
  cognitive scores

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosugery, Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No